CLINICAL TRIAL: NCT05986708
Title: The Effect of Guided Self-Determination (GSD) Method on Treatment Adherence, Fluid Control, Self-Efficancy, Anxiety and Quality of Life in Patients Undergoing Hemodialysis
Brief Title: Application of Guided Self- Determination (GSD) Method in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fusun Uzgor, research assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EskisehirOsmangaziU
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hemodialysis Patients
Keywords: guided self-determintion; hemodialysis; treatment adherence; quality of life; fluid control; anxiety
MeSH Terms: conditions — Treatment Adherence and Compliance; Anxiety Disorders | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The intervention group conducted 6 sessions of interviews with the researcher using the worksheets within the scope of the guided self-determination method.
  Interventions: Other: interview
- control (No Intervention): No intervention was made to the individuals in the control group.

INTERVENTIONS:
Other: interview — In addition to routine treatment and care, the patients in the application group were interviewed by the researcher once a week for 6 weeks, within the first hour of HD treatment, for a total of 6 sessions, each session being approximately 30 minutes-1 hour, within the scope of the guided self-determination method.
  Arms: intervention

SUMMARY:
The aim of this study is to assess how guided self-determination method affects adherence to treatment, fluid control, self-efficacy, anxiety level and quality of life in hemodialysis patients.

The population of the study consisted of patients who received HD treatment at Private Eskişehir Anatolian Dialysis Center and Eskişehir Osmangazi University Health, Practice and Research Hospital Dialysis Unit between April 2022 and October 2022. The sample of the study was 65 patients who met the inclusion criteria in the specified population.

Individual Identification Form, Biological/Biochemical Data Form, End Stage Renal Failure Compliance Scale, Hemodialysis Patients Fluid Control Scale, General Self-Efficacy Scale, Beck Anxiety Scale and SF-36 Quality of Life Scale Short Form were used to collect research data.

DETAILED DESCRIPTION:
Guided Self- Determination (GSD) is a self-management support intervention aimed at supporting decision making and problem solving and helping patients suffering from a chronic disease to improve their life skills. GSD aims to support and develop the self management ability of the patients' chronic illness according to their own needs and desires by sharing psychosocial aspects, enabling active involvement of the patient in goal setting and treatment decisions, and thus developing positive autonomy and responsibility in the patient. This method is based on the idea that there is a potential for change in the patient-nurse relationship to support mutual understanding and cooperation.

This method consists of interviews using structured self-evaluation forms based on theories. It aims to guide the patient to gain skills for self-determination and self management by using these self-evaluation forms in thinking, goal setting, and problem solving .The self-assessment forms include four themes: the patient-healthcare professional relationship, illness and life, the relationship between ideal and reality, and working for change. The aim is to guide patients and healthcare professionals through mutual thinking using a six-step interaction process. These six stages are (i) establishing a clear mutual patient-nurse relationship (ii) self-discovery, (iii) self-understanding, (iv) shared decision making, (v) action, and (vi) feedback from action. In each interview, the patient fills out the self-evaluation forms in advance to encourage sharing before and during the interview with the nurses.

In our study, there are 2 groups; intervention and control groups. In addition to routine treatment and care, the patients in the intervention group were interviewed by the researcher once a week for 6 weeks, with a total of 6 sessions of directed self-determination, each session being approximately 30 min-1 hour before HD treatment. The interview time was determined in consultation with the patients, and when the patient forgot/missed an interview, he was offered an appointment for another interview if he wanted to continue the study. Evaluations of the patients in both groups was performed with biological and/or biochemical data, ESRD-SQ, General Self-Efficacy Scale, HHSSK, SF-36 Quality of Life Scale Short Form and the Beck Anxiety Scale at the end of the interviews (week 6) and week 18, conducted within the scope of guided self-determination method.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70,
* Literate,
* Having end-stage renal failure,
* Receiving HD treatment,
* Able to communicate in Turkish,
* No hearing or vision loss,
* Conscious Open,
* Patients who volunteer to participate in the study.

Exclusion Criteria:

* End-stage renal failure hospitalized due to emergency,
* Receiving HD treatment for a reason other than end-stage renal disease,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The change in treatment adherence in hemodialysis patients | week 0, week 6, and week 18 of the study
  Treatment adherence was evaluated in study with the End Stage Kidney Disease Adherence Scale (ESRD-AQ) .The End Stage Kidney Disease Adherence Scale evaluates patients' participation in hemodialysis treatment, their medication use, their adherence with fluid restriction and diet.
  The validity and reliability analysis of the scale was made on 9 items. The total score that can be obtained from the scale varies between 0-1200. As the score obtained from the scale increases, the level of adherence to treatment increases.
The change in fluid control in hemordialysis patients | week 0, week 6, and week 18 of the study
  Fluid control was evaluated with "Fluid Control in Hemodialysis Patients Scale". This scale has a total of 24 items and three sub-dimensions. Information sub-dimension: 1.-7. from questions; behavior sub-dimension 8.-18. From the questions; attitude sub-dimension 19.-24. consists of questions. The lowest score obtained from the scale is 24, the highest score is 72, and as the score increases, patients' compliance with fluid control increases.
The change in self-efficancy in hemodialysis patients | week 0, week 6, and week 18 of the study
  Self-efficancy was evaluated at 0th week, 6th weeks and 18th weeks in study with General Self-Efficancy Scale".This scale has a total of 24 items. Each of the 10 items in the scale receives scores ranging from 1 to 4. The lowest score obtained from the scale is evaluated as 10 and the highest score as 40, and as the scale score increases, the self-efficacy score increases.
The change in quality of life in hemodialysis patients | week 0, week 6, and week 18 of the study
  The change in quality of life in hemodialysis patients was evaluated with the Short Form of the Quality of Life Scale (SF 36). The scale consists of 36 questions and the last four weeks of the individuals are questioned. The scale consists of eight sub-dimensions and the sub-dimensions is evaluated separately. On the scale, "0" indicates poor health, "100" indicates good health.
The change in anxiety level in hemodialysis patients | week 0, week 6, and week 18 of the study
  Anxiety level was evaluated with Beck Anxiety Inventory. It is a self-assessment scale consisting of 21 items and scored between 0-3. With the questions asked to the person, it is questioned to what extent the feeling of distress has disturbed him in the last week. Scores from the scale range from 0 to 63, with 8-15 points = mild anxiety, 16-25 points = moderate anxiety, 26-63 points = severe anxiety.

SECONDARY OUTCOMES:
The change in intradialytic weight (kg) in hemodialysis patients | week 0, week 6, and week 18 of the study
  Interdialytic weight was measured by the weight difference between two hemodialysis sessions.
The change in serum potassium (mEq/L) value in hemodialysis patients | week 0, week 6, and week 18 of the study
  Serum potassium value was taken from the patient file. Normal serum potassium is 3.5 to 5.5 mEq/L.
The change in serum phosphorus (mmol/L) value in hemodialysis patients | week 0, week 6, and week 18 of the study
  Serum phosphorus value was taken from the patient file. Normal serum phosphorus value is 3.5 to 5.5 mmol/L.
The change in serum calcium (mg/dl) in hemodialysis patients | week 0, week 6, and week 18 of the study
  Serum calcium value was taken from the patient file. Normal serum calcium value is 8.6 to 10.0 mg/dl.
The change in serum albumin (g/dl) in hemodialysis patients | week 0, week 6, and week 18 of the study
  Serum calcium value was taken from the patient file. Normal serum albumin value is 3.4 to 4.8 g/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Füsun Uzgör, Principal Investigator — eskişehir osmangazi university
Locations (1):
- Eskişehir Osmangazi University Faculty of Health Sciences, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No